CLINICAL TRIAL: NCT03042481
Title: Comparison and Prediction of Off-therapy Response in Patients of Chronic Hepatitis B Treated With Entecavir or Tenofovir and Achieved Criteria of Stopping Therapy by APASL Guideline
Brief Title: Off-therapy Response After Stopping Entecavir or Tenofovir
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-G(I)-20160015
Record Dates: First submitted 2017-01-23; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis B; entecavir; tenofovir; off-therapy; relapse
MeSH Terms: conditions — Hepatitis B, Chronic; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Pegylated-interferon (Peg-IFN) α-2a, entecavir (ETV) and tenofovir disoproxil fumarate (TDF) are current recommended first-line antiviral therapies for chronic hepatitis B (CHB). Compared with Peg-IFN therapy, nucleot(s)ide analogue (NUC) therapy has the advantages of having a potent antiviral effect, and good tolerance without side effect. The long-term safety and efficacy of ETV and TDF therapy had also been identified. However, poor durability of the effectiveness after stopping NUC therapy are encountered in the majority of patients. Previous study identified a high HBV relapse rate of over 50% in HBeAg- positive CHB patients treated with lamivudine. A recent study investigating the post-treatment durability of ETV showed that higher to 45.3% of the HBeAg-negative CHB patients happened a clinical relapse within 1-year after stopping ETV therapy. TDF is another recommended first line NUC with high potency and high genetic barrier. Although the efficacy of long-term TDF therapy had been identified, there is lack of data regarding the off-therapy response in CHB patients with TDF therapy currently. Only a small scale of patients treated with TDF were included in a recent study investigating off-therapy relapse in non-cirrhotic HBeAg-negative CHB patients after greater than 4 years of NUC therapy. In addition, the factors associated with off-therapy response are also still uncertain.

The investigators plan to enrolled 400 CHB patients who had received oral antiviral therapy ETV or TDF and achieved the Asia Pacific association of the study of liver (APASL) criteria of stopping NUC therapy. The aims of the study are to investigate the rate of HBV relapse including virological and clinical relapse in all and between patients with ETV and TDF therapy, and to identify the predictive factors of relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients >20 years of age
2. Positive HBsAg for more than 6 months prior to ETV or TDF therapy.
3. HBV DNA ≥20,000 IU/mL and alanine aminotransferase (ALT) levels ≥ 2 fold the upper limit of normal (ULN) for the HBeAg-positive patients, and HBV DNA ≥2000 IU/mL and ALT levels ≥ 2 fold the ULN for the HBeAg-negative patients prior to ETV or TDF therapy.
4. Achieve the APASL criteria of stopping NUC therapy including HBeAg seroconversion (negative HBeAg and positive HBeAb) with HBV DNA loss measured at two consecutive occasions at least 6 months apart for HBeAg positive patients; more than 2 years therapy with undetectable HBV DNA documented on three separate occasions 6 months apart for HBeAg negative patients.

Exclusion Criteria:

1. Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) co-infection.
2. History or other evidence of a medical condition associated with chronic liver disease other than CHB (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
3. Evidence of drug abuse (including excessive alcohol consumption).
4. Prophylactic use of ETV or TDF therapy. (for cancer chemotherapy or post-transplant immunosuppressive therapy prophylaxis)
5. Patients who have clinical evidence of liver cirrhosis.
6. Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHB patients who had received oral antiviral therapy ETV or TDF and achieved the Asia Pacific association of the study of liver (APASL) criteria of stopping nucleot(s)ide therapy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Rate of HBV relapse | One year after stopping HBV antiviral therapy
Rate of HBV relapse | Two year after stopping HBV antiviral therapy

SECONDARY OUTCOMES:
Rate of severe hepatitis flare (ALT level ≥10 fold the ULN) with/without hepatic decompensation (total bilirubin ≥2). | One year after stopping NUCs
Rate of severe hepatitis flare (ALT level ≥10 fold the ULN) with/without hepatic decompensation (total bilirubin ≥2). | Two year after stopping HBV antiviral therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hepatobiliary, Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan